CLINICAL TRIAL: NCT07116811
Title: The Effect of Steroids Treatment for Facial Nerve Function Protection in Post-surgical Vestibular Schwannoma Patients (SAF-NRVS): a Multicenter, Randomized, Double-blind, Placebo-parallel Controlled Trial
Brief Title: Steroids for Facial Nerve Function Protection in Post-surgical Vestibular Schwannoma Patients
Acronym: SAF-NRVS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Wang Jia, Professor of Beijing Tiantan Hospital, Capital Medical University, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2025-137-02
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Vestibular Schwannoma; Facial Nerve Paralysis
Keywords: Steroids; Facial Nerve Function; Intraoperative Neurophysiological Monitoring; Randomized Controlled Trial; Facial Palsy
MeSH Terms: conditions — Neuroma, Acoustic; Bell Palsy; Facial Paralysis

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. Patients with untreated unilateral vestibular schwannoma and good preoperative facial nerve function will be randomized in a 1:1 ratio to receive either steroid therapy or placebo. All participants will undergo craniotomy with intraoperative neurophysiological monitoring to ensure adequate facial nerve function preservation. Treatment will be initiated on the day of surgery and continued for 10 days. The primary outcome is the proportion of patients with good facial nerve recovery at 90 days postoperatively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study adopted a double-blind design. Study drugs and placebos are identically packaged. The dosage form, size, color, weight, smell, and taste of the placebo were basically similar to those of the research drug, and there was no risk of blinding. Personnel involved in randomization or potentially exposed to treatment allocation (including pharmacy staff) are not involved in patient care, outcome assessment, or data analysis. Blinded investigators and outcome assessors remain unaware of treatment assignments throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroids Group (Experimental): Methylprednisolone sodium succinate (80 mg/day) on days 1-3 post-surgery, followed by prednisone acetate (20 mg/day) on days 4-10.
  Interventions: Drug: Steroids therapy
- Placebo Group (Placebo Comparator): Methylprednisolone sodium succinate placebo on days 1-3 post-surgery, followed by prednisone acetate placebo on days 4-10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Steroids therapy — Methylprednisolone sodium succinate 80 mg powder dissolved in 100 mL of sodium chloride solution (intravenous infusion, once daily) from the day of surgery to day 3, followed by 20 mg of prednisone acetate (oral intake, once daily) from day 4 to day 10.
  Arms: Steroids Group
Drug: Placebo — Methylprednisolone sodium succinate placebo powder dissolved in 100 mL of sodium chloride solution (intravenous infusion, once daily) from the day of surgery to day 3, followed by prednisone acetate placebo (oral intake, once daily) from day 4 to day 10.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of steroids treatment compared with placebo in preserving facial nerve function after craniotomy in patients with vestibular schwannoma who have not received preoperative treatment and have good intraoperative facial nerve function.

DETAILED DESCRIPTION:
Vestibular schwannoma (VS) is a benign tumor arising from the vestibular nerve. Surgical resection is a common treatment, and intraoperative neurophysiological monitoring (IONM) is widely used to protect facial nerve function. However, postoperative facial nerve paralysis remains a common complication, affecting patients' appearance, confidence, and quality of life.

Steroids are often used to reduce inflammation and edema in idiopathic facial palsy, but their efficacy and safety in post-surgical VS patients remain uncertain. The mechanism of post-surgical facial nerve dysfunction is more complex than idiopathic palsy and may involve physical traction, vascular compromise, or inflammatory injury.

This study (SAF-NRVS) is a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. Patients aged 18 to 60 years with a clinically confirmed untreated unilateral vestibular schwannoma will be enrolled. Eligible patients must have no preoperative facial paralysis (grade I according to the House-Brackmann grading system), and have good intraoperative facial nerve function as determined by intraoperative neurophysiological monitoring. Participants will be randomly divided into two groups in a 1:1 ratio. Intervention group (Steroids group) will receive 80 mg of methylprednisolone sodium succinate powder dissolved in 100 ml of sodium chloride (NaCl) solution by intravenous infusion once daily from the day of surgery to day 3, followed by 20 mg of prednisone acetate oral intake once daily from day 4 to day 10. Control group (Placebo group) will receive methylprednisolone sodium succinate placebo powder dissolved in 100 ml of NaCl solution by intravenous infusion once daily from the day of surgery to day 3, followed by prednisone acetate placebo oral intake once daily from day 4 to day 10. The primary outcome measure is the proportion of patients with good facial nerve function recovery at 90 days after surgery, defined as grade 1 or 2 according to House-Brackmann grading system.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years
2. Diagnosed with untreated unilateral vestibular schwannoma
3. No facial palsy before surgery (House-Brackmann grade I)
4. Intraoperative neurophysiological monitoring confirms good facial nerve function preservation, defined as: a）Post-tumor resection, evoked compound muscle action potential amplitude >420 μV under 0.05 mA stimulation；and b）The amplitude is >60% of baseline value measured before dural opening
5. Signed informed consent

Exclusion Criteria:

1. Contraindications for craniotomy
2. Patients requiring corticosteroids during the perioperative period, or with known corticosteroid contraindications
3. Patients or first-degree relatives with a confirmed diagnosis of neurofibromatosis type 2 (NF2)
4. Karnofsky Performance Status (KPS) score <90 before disease onset
5. Pregnant or planning to become pregnant during the study period
6. Participation in other interventional clinical trials
7. Judged unsuitable by the investigators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 364 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Good facial nerve function (House-Brackmann grade I or II) at 90 days after surgery | at 90 (±7) days after surgery
  Defined as House-Brackmann grade I or II.

SECONDARY OUTCOMES:
Good facial nerve function (House-Brackmann grade I or II) at 10 days after surgery | at 10 days after surgery
  Defined as House-Brackmann grade I or II.
Complete facial nerve function recovery (House-Brackmann grade I) at 90 days after surgery | at 90 (±7) days after surgery
  Defined as House-Brackmann grade I
Complete facial nerve function recovery (House-Brackmann grade I) at 10 days after surgery | at 10 days after surgery
  Defined as House-Brackmann grade I
Complete facial nerve function recovery (Sunnybrook scale 100 score) at 90 days after surgery | at 90 (±7) days after surgery
  Sunnybrook Facial Grading System will be used. Score of 100 represents complete recovery.
Complete facial nerve function recovery (Sunnybrook scale 100 score) at 10 days after surgery | at 10 days after surgery
  Sunnybrook Facial Grading System will be used. Score of 100 represents complete recovery.
Adverse events within 90 days | Within 90 (±7) days after surgery
Serious adverse events within 90 days | Within 90 (±7) days after surgery
Adverse events within 10 days | Within 10 days after surgery
Serious adverse events within 10 days | Within 10 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No